CLINICAL TRIAL: NCT04367311
Title: A Phase II Study of Adjuvant Treatment With Cisplatin-based Chemotherapy Plus Concomitant Atezolizumab in Patients With Stage I (Tumors ≥ 4cm), IIA, IIB, and Select Stage III [Any T1-3 N1-2 and T4N0-2] Resected Non-small Cell Lung Cancer (NSCLC) and the Clearance of Circulating Tumor DNA (ctDNA) Big Ten Cancer Research Consortium BTCRC-LUN19-396
Brief Title: Adjuvant Treatment With Cisplatin-based Chemotherapy Plus Concomitant Atezolizumab in Patients With Stage I (Tumors ≥ 4cm), IIA, IIB, and Select Stage III [Any T1-3 N1-2 and T4N0-2] Resected Non-small Cell Lung Cancer (NSCLC) and the Clearance of Circulating Tumor DNA (ctDNA)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nasser Hanna (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nasser Hanna, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-LUN19-396
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — atezolizumab; Docetaxel; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSC: Non-squamous cell tumors (Experimental): Atezolizumab 1200mg, Pemetrexed 500 mg/m^2, Cisplatin 60-75 mg/m^2
  Interventions: Drug: Atezolizumab; Drug: Cisplatin; Drug: Pemetrexed
- SC: Squamous cell tumors (Experimental): Atezolizumab 1200mg, Docetaxel 60-75 mg/m^2, Cisplatin 60-75 mg/m^2
  Interventions: Drug: Atezolizumab; Drug: Docetaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg
Drug: Docetaxel — Docetaxel 60-75 mg/m^2
  Arms: SC: Squamous cell tumors
Drug: Cisplatin — 60-75 mg/m^2
Drug: Pemetrexed — Pemetrexed 500mg/m^2
  Arms: NSC: Non-squamous cell tumors

SUMMARY:
The vast majority of patients with stage I (tumors ≥ 4cm), IIA, IIB (and select stage III) NSCLC are managed with upfront surgery, followed by adjuvant chemotherapy. However, relapse rates remain high and are primarily due to distant, metastatic disease. Previous meta-analysis evaluating the use of neo-adjuvant chemotherapy and adjuvant chemotherapy demonstrate a similar impact on improved disease free survival (DFS) and overall survival (OS). The role of checkpoint inhibitors has been proven to be effective in the treatment of patients with advanced NSCLC, regardless of histology and PD-L1 expression. Results from trials evaluating the use of checkpoint inhibitors alone or in combination with chemotherapy in the neoadjuvant setting for early stage disease are promising. However, there are no trials evaluating the role of concomitant chemotherapy and checkpoint inhibitors in the adjuvant setting. In addition, emerging data supports the use of ctDNA as a promising biomarker for early detection of minimal residual disease and have indicated that the presence of detectable ctDNA after surgery for localized lung cancer is correlated with a 90-100% chance for disease recurrence. Therefore, we propose this current study assessing concomitant chemotherapy plus Atezolizumab in the adjuvant setting for patients with stage I (tumors ≥ 4cm), IIA, IIB (and select stage III) NSCLC who have detectable ctDNA after surgery. The clearance of ctDNA will serve as a surrogate for long term DFS and OS in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age >= 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 28 days prior to registration.
* Patients must have undergone complete surgical resection of their stage I (tumors >= 4cm), IIA, IIB, and select stage III [any T1-3 N1-2 and T4N0-2] NSCLC according to the AJCC 8th edition with negative margins (R0).
* Squamous or non-squamous NSCLC histology. Cancers with a histology of "adenosquamous" are considered a type of adenocarcinoma and thus "non-squamous histology".
* Surgery for this lung cancer must be completed <= 60 days prior to starting treatment.
* Must have tissue available to perform prospective correlative testing. Tissue block is preferred but 10-15 unstained slides (5 μm thick) are also acceptable. If prior PD-L1 results with Dako 22C3 antibody are not available, an additional 5 unstained slides (4 μm thick) must be submitted.
* Demonstrate adequate organ function as defined in the protocol; all screening labs to be obtained within 28 days prior to registration.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

  * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of atezolizumab.
  * A woman is considered of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (> or equal to 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Contraception method must begin starting from the time of informed consent until 5 months after treatment discontinuation.
* For men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 5 months after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

* Tumors that have any component of small cell or large cell neuroendocrine histology are NOT eligible.
* Tumors that are known to harbor EGFR mutations or ALK re-arrangements are NOT eligible.
* Prior chemotherapy, radiation therapy, or immunotherapy is NOT allowed for the treatment of this lung cancer.
* Prior chemotherapy and/or radiation therapy is permissible for the treatment of other previous cancers, but must have been completed at least 3 months prior to registration for this trial.
* Other active cancers.
* History of leptomeningeal disease.
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 1 week prior to registration.
* Has severe hypersensitivity (>= Grade 3) to atezolizumab and/or any of its excipients.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or infusion proteins.
* Has active or history of autoimmune disease or immune deficiency that includes but is not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis.
* Known interstitial lung disease that is symptomatic or may interfere with detection or management of suspected drug-related pulmonary toxicity are not permitted.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g. PleurX) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12mg/dL or corrected serum calcium >ULN).
* Significant cardiovascular disease within 3 months prior to initiation of study treatment (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident), unstable arrhythmia, or unstable angina.
* For patients receiving therapeutic anticoagulation: unstable anticoagulant regimen.
* Has a severe infection within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Has a known history of Human Immunodeficiency Virus (HIV). Note: HIV testing is not required.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection. Note: If Hepatitis B and Hepatitis C status is unknown, testing is required:

  * Subject must have negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. The HBV DNA test will be performed only for patients who have a positive total HBcAb test.
  * Subject must have negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test. A positive HCV RNA test is sufficient to diagnose active HCV infection in the absence of an HCV antibody test.
* Has a known history of active TB (Bacillus Tuberculosis).
* Prior allogeneic stem cell or solid organ transplantation.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 5 months after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with undetectable ctDNA after 4 cycles of adjuvant chemotherapy + Atezolizumab plus up to 13 additional cycles of Atezolizumab in patients with stage I (tumors ≥ 4cm), IIA, IIB, and select stage III [any T1-3 N1-2 and T4N0-2] | Up to 17 cycles (13 months)
  To estimate the percentage of patients with undetectable circulating tumor DNA (ctDNA) after 4 cycles of adjuvant chemotherapy + Atezolizumab plus up to 13 additional cycles of Atezolizumab in patients with stage I (tumors ≥ 4cm), IIA, IIB, and select stage III [any T1-3 N1-2 and T4N0-2] NSCLC who have detectable ctDNA after surgery, but prior to adjuvant therapy.
  At each time point, ctDNA detection status (detectable or not detectable) will be determined by CAPP-seq using the Monte Carlo-based ctDNA detection index cutoff point of < 0.05, as described by Newman et al [53, 54]. If ctDNA detection index is > 0.05, ctDNA will be classified as not detected at that time point, whereas if < 0.05 then it will be classified as detected.

SECONDARY OUTCOMES:
Percentage of patients with clearance of ctDNA after 4 cycles of adjuvant chemotherapy + Atezolizumab | 4 cycles (3 months)
  To estimate the percentage of patients with clearance of ctDNA after 4 cycles of adjuvant chemotherapy + Atezolizumab in patients with stage I (tumors ≥ 4 cm), IIA, IIB, and select stage III [any T1-3 N1-2 and T4N0-2] NSCLC who have undergone surgical resection with detectable ctDNA after surgery.
Percentage of patients with clearance of ctDNA after 8 cycles (4 cycles of adjuvant chemotherapy + Atezolizumab plus 4 additional cycles of Atezolizumab) | 8 cycles (6 months)
  To estimate the percentage of patients with clearance of ctDNA after 8 cycles (4 cycles of adjuvant chemotherapy + Atezolizumab plus 4 additional cycles of Atezolizumab) in patients with stage I (tumors ≥ 4 cm), IIA, IIB, and select stage III [any T1-3 N1-2 and T4N0-2] NSCLC who have undergone surgical resection with detectable ctDNA after surgery.
Percentage of patients with clearance of ctDNA after 12 cycles (4 cycles of adjuvant chemotherapy + Atezolizumab plus 8 additional cycles of Atezolizumab) | 12 cycles (9 months)
  To estimate the percentage of patients with clearance of ctDNA after 12 cycles (4 cycles of adjuvant chemotherapy + Atezolizumab plus 8 additional cycles of Atezolizumab) in patients with stage I (tumors ≥ 4 cm), IIA, IIB, and select stage III [any T1-3 N1-2 and T4N0-2] NSCLC who have undergone surgical resection with detectable ctDNA after surgery.
Percentage of patients with clearance of ctDNA during or after adjuvant chemotherapy + Atezolizumab followed by Atezolizumab for up to 13 additional cycles who had no detectable ctDNA after surgery | Up to 17 cycles (13 months)
  To estimate the percentage of patients with clearance of ctDNA during or after adjuvant chemotherapy + Atezolizumab followed by Atezolizumab for up to 13 additional cycles who had no detectable ctDNA after surgery
Percentage of pts with clearance of ctDNA after 4 cycles of adj. chemotherapy + Atezolizumab plus up to 13 additional cycles of Atezolizumab | Up to 17 cycles (13 months)
  To estimate the percentage of patients with undetectable ctDNA after 4 cycles of adjuvant chemotherapy + Atezolizumab plus up to 13 additional cycles of Atezolizumab in patients with stage I (tumors ≥ 4 cm), IIA, IIB, and select stage III [any T1-3 N1-2 and T4N0-2] NSCLC who have undergone surgical resection, regardless of ctDNA status after surgery
1 year Disease Free Survival (DFS) in all patients | 1 year
  To estimate the 1 year Disease Free Survival (DFS) in all patients treated on study
1 year Disease Free Survival (DFS) in patients with no detectable ctDNA after 4 cycles of adjuvant chemotherapy + Atezolizumab who had detectable ctDNA after surgery. | 1 year
  To estimate the 1 year Disease Free Survival (DFS) in patients with no detectable ctDNA after 4 cycles of adjuvant chemotherapy + Atezolizumab who had detectable ctDNA after surgery.
1 year Disease Free Survival (DFS) in patients with detectable ctDNA after 1 year of adjuvant therapy on study | 1 year
  1 year Disease Free Survival (DFS) in patients with detectable ctDNA after 1 year of adjuvant therapy on study

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, MD, Principal Investigator — Indiana University
Locations (9):
- United States (9):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Summit Health, Berkeley Heights, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University Clinical Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No